CLINICAL TRIAL: NCT00688961
Title: A Pilot Study of the Effects of Omacor (Alone and With Aspirin) on Platelet Function in Healthy Subjects
Brief Title: Effects of Omacor and Aspirin on Platelet Function
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sanford Research (Other)
Responsible Party: William S. Harris, Sanford Research/USD
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: WSH-001
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: omega-3 fatty acids; aspirin; platelet aggregation; Healthy volunteers; no disease
MeSH Terms: interventions — Aspirin; Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (No Intervention): Baseline
- 2 (Experimental): Aspirin (1 day after a single, 625 mg dose)
  Interventions: Drug: Aspirin
- 3 (Experimental): Omacor
  Interventions: Drug: omega-3 acid ethyl esters
- 4 (Experimental): Omacor plus aspirin
  Interventions: Drug: Aspirin; Drug: omega-3 acid ethyl esters

INTERVENTIONS:
Drug: Aspirin — generic aspirin
  Arms: 2; 4
Drug: omega-3 acid ethyl esters — 4, 1 g capsules q.d.
  Other Names: Omacor; Lovaza
  Arms: 3; 4

SUMMARY:
Omacor (now Lovaza) is a pharmaceutical omega-3 fatty acid product. Omega-3 fatty acids can affect blood clotting by altering the function of the blood platelets. Aspirin can do the same. The purpose of this study is to determine the individual and combined effects of these two agents on platelet function using a whole blood method.

DETAILED DESCRIPTION:
Overview

This study will explore the effects of 4 g/d of Omacor in healthy volunteers both with and without concomitant aspirin therapy. The study will utilize three different analytical approaches to assess platelet activation and function.

Objective

The purpose of this exploratory study is to gather preliminary information on the effects of Omacor on a platelet function in healthy volunteers, both with and without concomitant aspirin therapy, in order to lay the groundwork for future studies in cardiac patients taking Omacor in combination with aspirin and clopidogrel.

Background/Significance

Omacor (omega-3 fatty acid ethyl esters) is approved for treatment of severe hypertriglyceridemia, and may soon be approved for the treatment of moderate hypertriglyceridemia in combination with statins. In other words, the use of Omacor will continue to expand. The package insert notes that physicians should be attuned to the possibility of increased bleeding tendencies with high dose (4 g/d) Omacor use despite the fact that clinically significant bleeding has virtually never been reported with this dose (or even up to 7 g of EPA+DHA) in studies in patients on concomitant anti-platelet therapy undergoing highly invasive vascular procedures (e.g., diagnostic catheterization, angioplasty, coronary artery bypass grafting). Nevertheless, because omega-3 fatty acids are known to inhibit platelet function and to increase bleeding times(1), it is prudent to explore and carefully define the effects of this dose of Omacor on platelet composition and function.

Primary and Secondary Endpoints

The primary endpoint will be the effects of Omacor ± aspirin on platelet aggregation measured by whole blood impedence aggregometry in Harris's laboratory.

The secondary aims are to explore some of the molecular mechanisms by which omega-3 fatty acids and/or aspirin may alter platelet function. These include spreading assays, and tests of calcium and ATP release (described below). Even if the whole blood aggregation assays are not altered by Omacor treatment (they will be altered by aspirin treatment), these tests are sensitive to more subtle alterations in platelet function that could be missed in platelet aggregation assays. Alternatively, omega-3 FAs could impact two independent pathways in opposite directions, resulting in a cancelling out of the overall effect on platelet aggregation. These more focused experiments will be conducted at Dr. Mark Larson's laboratory at Augustana College.

Experimental Design and Methodology

Design This will be an open-label, pre- and post, 4-week trial. Blood will be drawn on day 1 (baseline), day 2 (1 day after taking 650 mg of aspirin), day 29 (after taking Omacor for 28 days), and day 30 (Omacor + 650 mg of aspirin). Platelet aggregation will be tested in each blood sample.

Subjects Ten healthy volunteers will be recruited from among the staff of Sanford Research/USD, Sanford School of Medicine, and Sanford Hospital; patients, students, visitors, and subordinates of the investigators will not be eligible. Subjects may be male or female and between the ages of 21 and 60, non-smokers, and taking no medications, vitamin pills, nutritional supplements or herbal preparations. Subjects may not have a history of allergic reactions to aspirin, fish or fish oils. Birth control pills are not allowed. Subject cannot have an allergy to aspirin or to non-steroidal anti-inflammatory drug (NSAID) such as ibuprofen (Motrin, Advil, others), naproxen (Aleve, Naprosyn, Anaprox, others), indomethacin (Indocin), or ketoprofen (Orudis KT, Orudis, Oruvail), nabumetone (Relafen), oxaprozin (Daypro), or tartrazine. Other exclusions include: drinking more than three alcoholic beverages a day, or having any of the following conditions: an ulcer or bleeding in the stomach, liver or kidney disease, bleeding or blood clotting disorder (e.g., hemophilia), congestive heart failure, fluid retention, heart disease, high blood pressure, gout, asthma, arthritis, or nasal polyps.

Laboratory Methods Blood will be drawn into sodium citrate for all tests. Three agonists will be used in the whole blood aggregometry tests: thrombin, collagen and ADP(3). The output of this instrument (Chronolog Whole Blood Aggregometer, model 504) is in ohms, with higher impedance values indicating greater platelet aggregation. Because this test is conducted in whole blood (i.e., erythrocytes present), it is thought to be the most physiologically-relevant method for testing platelet function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be male or female and between the ages of 21 and 60,
* Non-smokers,
* Taking no medications, vitamin pills, nutritional supplements or herbal preparations.

Exclusion Criteria:

* Subjects may not have a history of allergic reactions to aspirin, fish or fish oils.
* Birth control pills are not allowed.
* Subject cannot have an allergy to aspirin or to non-steroidal anti-inflammatory drug (NSAID) such as ibuprofen (Motrin, Advil, others), naproxen (Aleve, Naprosyn, Anaprox, others), indomethacin (Indocin), or ketoprofen (Orudis KT, Orudis, Oruvail), nabumetone (Relafen), oxaprozin (Daypro), or tartrazine.
* Drinking more than three alcoholic beverages a day
* Having any of the following conditions:

  * an ulcer or bleeding in the stomach,
  * liver or kidney disease,
  * bleeding or blood clotting disorder (e.g., hemophilia),
  * congestive heart failure,
  * fluid retention,
  * heart disease,
  * high blood pressure,
  * gout,
  * asthma,
  * arthritis, or
  * nasal polyps.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Whole blood aggregometry in response to 4 agonists | Day 1, 2, 29, and 30

CONTACTS AND LOCATIONS:
Locations (1):
- Sanford Research/USD, Sioux Falls, South Dakota, United States